CLINICAL TRIAL: NCT06582472
Title: Early Retinal Neurodegeneration As Risk Factor, Biomarker and Pharmacological Target of Diabetic Retinopathy
Acronym: 2022-12376008
Status: Recruiting | Type: Observational
Sponsor: IRCCS Ospedale San Raffaele (Other)
Responsible Party: Principal Investigator, Francesco Bandello, Principal Investigator, IRCCS Ospedale San Raffaele
Other Study IDs: PNRR-MAD-2022-12376008
Record Dates: First submitted 2024-08-26; First posted 2024-09-03 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: Diabetic Retinopathy; Diabetic Retinopathy Associated with Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetic Retinopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- cohort 1 (longitudinal study): This group will include patients affected by type 2 diabetes for less than 10 years and without signs of diabetic retinopathy, nephropathy, and neuropathy.
  Interventions: Procedure: Ophthalmological examination including imaging assessments; Procedure: confocal analysis of cornea; Procedure: Dynamic Vessel Analyzer (DVA); Procedure: tear sampling collection; Procedure: blood sampling collection
- cohort 2 (longitudinal study): healthy controls: subjects in good general health as evidenced by medical history without diagnosis of type 2 diabetes
  Interventions: Procedure: Ophthalmological examination including imaging assessments; Procedure: confocal analysis of cornea; Procedure: Dynamic Vessel Analyzer (DVA); Procedure: tear sampling collection; Procedure: blood sampling collection
- cohort 1 (cross sectional study): Patients with a diagnosis of type 2 diabetes for longer than 20 years without clinical signs of retinopathy and other diabetic complications
  Interventions: Procedure: Ophthalmological examination including imaging assessments; Procedure: confocal analysis of cornea; Procedure: Dynamic Vessel Analyzer (DVA); Procedure: tear sampling collection; Procedure: blood sampling collection
- cohort 2 (cross sectional study): Patients with a diagnosis of type 2 diabetes for longer than 20 years with clinical signs of retinopathy and other diabetic complications
  Interventions: Procedure: Ophthalmological examination including imaging assessments; Procedure: confocal analysis of cornea; Procedure: Dynamic Vessel Analyzer (DVA); Procedure: tear sampling collection; Procedure: blood sampling collection

INTERVENTIONS:
Procedure: Ophthalmological examination including imaging assessments — Ophthalmological examination including imaging assessments (SD-OCT, Spectral Domain Optical Coherence Tomography, a procedure to study and quantify possible retinal neurodegeneration and OCT-A, Optical coherence tomography angiography, a procedure to study and quantify possible retinal vascular abnormalities)
Procedure: confocal analysis of cornea — Confocal analysis of cornea: a procedure to study and quantify possible corneal nerve degeneration as a marker of involvement of diabetic neuropathy
Procedure: Dynamic Vessel Analyzer (DVA) — Dynamic Vessel Analyzer (DVA), a device that measures the response of retinal arteries and veins to a standardized stimulus (flickering light) allowing direct quantification of the inflammatory status of the retinal vasculature
Procedure: tear sampling collection — Collect and analyze tear samples to identify biomarkers in tears and at the endothelium of the ocular surface through impression conjunctival cytology and the quantitative/qualitative analysis of pro-inflammatory cytokines
Procedure: blood sampling collection — collection and analysis of blood samples to identify diabetic retinopathy biomarkers and early abnormalities of the vascular retinal system.

SUMMARY:
Despite the evidence that diabetic retinopathy (DR) remains the first cause of blindness among the working-age population, it lacks a specific preventive treatment. This is because early mechanisms leading to the development of DR have been, until recently, unknown. Recent studies have suggested that the early stages of DR could be preceded by neuronal abnormalities, in particular retinal ganglion cell death, coupled with widespread retinal inflammation. According to these studies, endothelial dysfunction and the development of microaneurysms, the classic hallmarks of DR, could be the consequence of these early abnormalities.

This project will aim to verify whether neurodegeneration could represent at the same time: 1) a risk factor for subsequent development of DR (this will be investigated through a follow-up study in type 2 diabetic patients free of diabetic retinopathy). 2) a biomarker of the complication (if so, patients with long-standing diabetes in the absence of retinopathy should show no signs of neurodegeneration).

DETAILED DESCRIPTION:
The project is centered on a clinical study aimed to clarify whether early, diabetes-driven neurodegeneration (something that has been demonstrated by several seminal studies) is related (possibly causative) to the subsequent development of DR (a concept that is presently far from being confirmed but that, in case, would probably pave the way to identify for the first time a treatment for this diabetic complication.

This project includes two substudies:

* LONGITUDINAL STUDY: the aim is to verify whether the presence of retinal neurodegeneration in type 2 diabetic patients without DR increases the risk of subsequent development of retinal microaneurisms, the classic first vascular sign of DR; will enroll 90 individuals affected by type 2 diabetes and 30 healthy controls. All the subjects will be recruited during the first 6 months of the study and followed for 24 months (baseline, month 6, month 12, month 18, and month 24).
* CROSS-SECTIONAL STUDY: the aim is to verify the clinical evidence of retinal neurodegeneration in patients with type 2 diabetes diagnosed over 20 years and with overt diabetic retinopathy, compared to patients with type 2 diabetes diagnosed for over 20 years but no signs of diabetic retinopathy. Will be enrolled 30 individuals affected by type 2 diabetes with a duration of disease longer than 20 years and no clinical signs of DR and 30 individuals affected by type 2 diabetes with a duration of disease longer than 20 years and DR of any stage. All the subjects will be recruited during the first 6 months of the study and subjected to only one visit to the site.

ELIGIBILITY:
Inclusion Criteria - Longitudinal study (patients):

1. Participant is willing and able to give informed consent for participation in the trial.
2. Male or Female, aged 40 - 80 years;
3. In good general health as evidenced by medical history or diagnosed with type 2 diabetes for less than 10 years without clinical signs of retinopathy and other diabetic complications;
4. HbA1c level 7% or greater;

Inclusion Criteria - Longitudinal study (healthy controls)

1. Participant is willing and able to give informed consent for participation in the trial;
2. Male or Female, aged 40 - 80 years;
3. In good general health as evidenced by medical history without diagnosis of type 2 diabetes;

Inclusion Criteria - Cross-sectional study

1. Participant is willing and able to give informed consent for participation in the trial;
2. Male or Female, aged 40 - 80 years;
3. Patient with a diagnosis of type 2 diabetes for longer than 20 years in the absence or presence of clinical signs of retinopathy and other diabetic complications;
4. HbA1c level 7% or greater.

Exclusion Criteria (longitudinal study and cross-sectional study)

An individual who meets any of the following criteria will be excluded from participation in this study:

1. retinal or systemic diseases other than diabetes;
2. hypertension (BP values greater than 140/90 mm Hg);
3. anemia (hematocrit less than 35%);
4. smoking;
5. laser treatment and pregnancy

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The longitudinal study will include 90 individuals affected by type 2 diabetes and 30 healthy controls.
  The cross-sectional study will include 30 individuals affected by type 2 diabetes with a duration of disease longer than 20 years and no clinical signs of DR and 30 individuals (matched for age, gender and duration of diabetes) affected by type 2 diabetes with a duration of disease longer than 20 years and DR of any stage (in absence of laser treatment).
Sampling Method: Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2023-09-29 (Actual); Primary Completion 2025-05-19 (Estimated); Study Completion 2025-05-19 (Estimated)

PRIMARY OUTCOMES:
imaging assessment (OCT, Optical coherence tomography; OCT-A, Optical Coherence Tomography Angiography and Dynamic Vessel Analyzer); confocal microscopy, blood sampling collection and conjunctival impression cytology | 24 months
  * Evaluation of changes in neuroretinal morphology by OCT (Optical coherence tomography), in the morphology of the retinal vascular component by OCT-A, and retinal blood perfusion due to the presence/absence of a light signal by Dynamic Vessel Analyzer);
  * identification of retinal neurodegeneration factors as possible biomarkers of diabetic retinopathy, using conjunctival impression cytology and quantum/qualitative analysis of pro-inflammatory cytokines in tears and plasma;
  * assessment of the appearance of signs of corneal nerve degeneration by confocal microscopy in patients with signs of overt retinal neurodegeneration.

SECONDARY OUTCOMES:
imaging assessment (OCT, Optical coherence tomography; OCT-A, Optical Coherence Tomography Angiography and Dynamic Vessel Analyzer); confocal microscopy, blood sampling collection and conjunctival impression cytology | 24 months
  * Evaluation of changes in neuroretinal morphology by OCT (Optical coherence tomography), in the morphology of the retinal vascular component by OCT-A, and retinal blood perfusion due to the presence/absence of a light signal by Dynamic Vessel Analyzer);
  * identification of retinal neurodegeneration factors as possible biomarkers of diabetic retinopathy, using conjunctival impression cytology and quantum/qualitative analysis of pro-inflammatory cytokines in tears and plasma;
  * assessment of the appearance of signs of corneal nerve degeneration by confocal microscopy in patients with signs of overt retinal neurodegeneration.

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Irccs Ospedale San Raffaele, Milan, Italy/milan
  - IRCCS Ospedale San Raffaele _O.U. Ophthalmology, Milan, Italy

IPD SHARING:
Plan to Share IPD: No